CLINICAL TRIAL: NCT04942145
Title: Behaviour, Anxiety Management, Personality Traits and Coping of Dental Patients Through Virtual Reality
Brief Title: Effect of Virtual Reality on Dental Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, full professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Dental virtual reality
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-07

CONDITIONS: Child Behavior Problem; Anxiety, Dental
Keywords: virtual reality; dental anxiety; behaviour; psychological factors
MeSH Terms: conditions — Anxiety Disorders; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Active Comparator): With virtual reality. In order to relate the following variables with the effectiveness in reducing dental anxiety.MDAS TEST (Modified Dental Anxiety Scale) FIS TEST (Facial Imagen Scale) Revised Neo Personality Test (NEO-FFI) Brief Cope Inventory, (coping strategies)
  Interventions: Device: virtual reality in dental patients
- Control Grooup (Experimental): Without virtual reality. In order to relate the following variables with the effectiveness in reducing dental anxiety.MDAS TEST (Modified Dental Anxiety Scale) FIS TEST (Facial Imagen Scale) Revised Neo Personality Test (NEO-FFI) Brief Cope Inventory, (coping strategies)
  Interventions: Device: virtual reality in dental patients

INTERVENTIONS:
Device: virtual reality in dental patients — The behavioral anxiety response of dental patients (with and without virtual reality) related to psychological factors is studied.
  Participants self-complete the questionnaires

SUMMARY:
Clinicians should appreciate the effectiveness of virtual reality (VR) headsets for managing both the anxiety and the behaviour of dental patients. The aim of this study was to assess the effectiveness of using a VR headset as a distraction for managing the anxiety and behaviour of patients during their dental treatment related to underlying psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with dental needs.
* Children with parental consent

Exclusion Criteria:

* patients with cognitive impairments

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Dental anxiety | 3 years
  MDAS TEST
Behaviour | 3 years
  FIS TEST
Personality traits | 3 years
  NEOFFI TEST
coping strategies | 3 years
  BRIEF COPE INVENTORY

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Clinica Odontológica de la Universidad de Salamanca, Salamanca
  - Javier Montero, Salamanca

IPD SHARING:
Plan to Share IPD: No